CLINICAL TRIAL: NCT00955240
Title: Phase II Nonrandomized Multicenter Study of the Impact of Radiochemotherapy (65 Gy + Cisplatin + 5FU) Combined With Cetuximab in Patients Presenting With Locally Advanced Anal Cancer
Brief Title: Radiation Therapy, Cisplatin, Fluorouracil, and Cetuximab in Treating Patients With Locally Advanced Anal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate toxicity
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000642638; FRE-FNCLCC-ACCORD-16-0708 (Other: LNCLCC); EU-20941 (Other: European union); 2007-007029-38 (EudraCT Number)
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Anal Cancer
Keywords: stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; squamous cell carcinoma of the anus
MeSH Terms: conditions — Anus Neoplasms | interventions — Cetuximab; Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin
Drug: fluorouracil
Other: laboratory biomarker analysis
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as fluorouracil and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving radiation therapy together with combination chemotherapy and cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying giving radiation therapy together with cisplatin, fluorouracil, and cetuximab to see how well it works in treating patients with locally advanced anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the objective response (complete and partial) 8 weeks after completion of study treatment comprising radiotherapy, chemotherapy (fluorouracil and cisplatin), and cetuximab followed by additional radiotherapy in patients with locally advanced anal cancer.

Secondary

* Evaluate colostomy-free survival.
* Evaluate the local control rate (objective response and stabilization) at 8 weeks.
* Evaluate relapse-free survival at 5 years.
* Evaluate the intermediate objective response at the end of week 5 of radiotherapy.
* Evaluate overall survival at 5 years.
* Evaluate the duration of response.
* Evaluate acute toxicities according to CTCAE v3.0.
* Evaluate late toxicities at 5 years according to CTCAE v3.0.
* Study the tumor markers associated with response (survival without relapse) and toxicity.
* Study the genotypes of Fc-receptor immunoglobulins (FCGR2A and FCGR3) and their association with skin toxicity, objective survival, and relapse-free survival.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV on days 0, 7, 14, 21, 28, and 35; fluorouracil IV on days 7-10 and 35-38; and cisplatin IV over 2 hours on days 7 and 35. Beginning on day 7, patients also undergo radiotherapy 5 days a week for 5 weeks (weeks 2-6). Two weeks after finishing this treatment, patients undergo additional radiotherapy* 5 days a week for 2 weeks (weeks 9 and 10).

NOTE: *Some patients may undergo brachytherapy.

Blood and tissue samples are collected for further analysis.

After completion of study treatment, patients are followed up for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed anal cancer

  * Squamous cell disease
  * Locally advanced, non-metastatic disease
  * One of the following clinical TNM stages:

    * T2, N0, M0 (largest diameter ≥ 3 cm)
    * T3-T4, N0, M0
    * Any T, N1-N3, M0
* No undifferentiated small cell carcinoma or adenocarcinoma
* Measurable disease according to RECIST criteria
* Undergone endorectal ultrasound or MRI to evaluate the primary tumor
* Undergone thoraco-abdomino-pelvic scan to evaluate tumor extension
* Disease suitable to receive radiotherapy and chemotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Leukocytes ≥ 4,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Creatinine clearance > 60 mL/min
* ALT and AST ≤ 5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Total bilirubin ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* No history of cancer within the past 8 years except for in situ cervical cancer or previously treated basal cell carcinoma of the skin
* No contraindications to any component of study therapy
* No serious uncontrolled illness
* No symptomatic grade 1 angina pectoris or angina pectoris ≥ grade 2
* No congestive heart failure
* No peripheral sensory neuropathy
* No uncontrolled diabetes
* No HIV positivity
* No geographical, social, or psychological situations that preclude medical follow up
* Affiliated with a social security system
* No patient deprived of liberty or under trusteeship

PRIOR CONCURRENT THERAPY:

* Patients with a diverting colostomy are eligible
* No prior excision of this tumor
* No prior chemotherapy or radiotherapy for the treatment of this cancer or any other history of radiotherapy or pelvic brachytherapy
* No concurrent coumarin anticoagulants, phenytoin, sorivudine or brivudine, antacids, or allopurinol
* Not registered in another clinical trial with an experimental drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2010-11-26 (Actual); Study Completion 2010-11-26 (Actual)

PRIMARY OUTCOMES:
Objective response (complete and partial) according to RECIST criteria at 8 weeks after completion of study treatment

SECONDARY OUTCOMES:
Survival rate at 3 and 5 years
Colostomy-free survival at 3 and 5 years
Duration of objective response

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deutsch, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (20):
- France (20):
  - Institut Bergonie, Bordeaux
  - CHU Hopital A. Morvan, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Hopital, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Charles Nicolle, Rouen
  - Centre Hospitalier Prive Saint-Gregoire, Saint-Grégoire
  - Clinique Du Parc, Toulouse
  - Groupe Oncorad Garonne, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif